CLINICAL TRIAL: NCT02188056
Title: Observational Prospectif Monocentric Registry of Patients Suffering From VIE
Acronym: REMOTEV
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 003-14
Record Dates: First submitted 2014-07-03; First posted 2014-07-11 (Estimated); Last update posted 2025-09-05 (Actual); Status verified 2014-07

CONDITIONS: Venous Thromboembolic Disease
Keywords: Venous; Thromboembolic; Pulmonary embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with an episode of VTE (DVT and / or PE) have a mortality rate of 16-21% at 1 year after diagnosis. Morbidity associated with VTE is marked by the risk of recurrence, estimated at 30% and estimated at 29% after 8 years of follow post-thrombotic syndrome. For a number of these patients, risk factors have been identified (congenital or acquired thrombophilia, cancer, postpartum, surgery, prolonged immobilization, etc..). In 25-50% of cases, the etiology remains unknown, justifying the need for well-conducted studies to determine other potential risk factors. In addition, the expansion of treatment options with the arrival on the market of new direct oral anticoagulants, allows comparative studies on the effectiveness and frequency of adverse events for each treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of venous thromboembolism established by a validated test (venous Doppler ultrasound of the lower limbs, pulmonary angiography, lung scan ventilation / perfusion),
* diagnosis of venous thromboembolism made within 15 days,
* the previous inclusion in the register (outpatient or inpatient)

Exclusion Criteria:

* person doesn't wish to participate in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with a venous thromboembolic event, hospitalized in the Department of Vascular Diseases and Hypertension, UF 1311 will included in the registry prospectively.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-10-01; Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
incidence of recurrent thromboembolic | at 1 year post-diagnosis
bleeding complications incidence | at 1 year post-diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Dominique STEPHAN, MD, PhD, Principal Investigator — Strasbourg University Hospital, France
Locations (1):
- Service Des Maladies Vasculaires - Hta - Nhc, Strasbourg, France